CLINICAL TRIAL: NCT02592954
Title: Effect of Broccoli Sprout Extract on Keratinocyte Differentiation in Normal Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: BSE2015
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Epidermolysis Bullosa Simplex; Pachyonychia Congenita
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Pachyonychia Congenita | interventions — jojoba wax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Jojoba oil with broccoli sprout extract (Experimental): 500nmol of broccoli sprout extract in 1ml of jojoba oil will be applied to the same arm every night under saran wrap for 1 week
  Interventions: Drug: Jojoba oil with broccoli sprout extract
- Jojoba oil (Placebo Comparator): 1ml of jojoba oil will be applied to the same arm every night under saran wrap for 1 week
  Interventions: Drug: Jojoba oil (placebo)

INTERVENTIONS:
Drug: Jojoba oil with broccoli sprout extract — 500nmol of broccoli sprout extract in 1ml of jojoba oil will be applied to the same arm every night under saran wrap for 1 week
  Arms: Jojoba oil with broccoli sprout extract
Drug: Jojoba oil (placebo) — 1ml of jojoba oil will be applied to the same arm every night under saran wrap for 1 week
  Arms: Jojoba oil

SUMMARY:
Adult participants will apply a broccoli sprout extract-jojoba oil compound to one arm every night under occlusion for 1 week. Jojoba oil alone will be applied to the other arm. At the end of 1 week, a 6mm punch biopsy will be taken from both arms and analyzed via polymerase chain reaction (PCR) and immunohistochemistry for differences in various skin proteins.

DETAILED DESCRIPTION:
10 adult volunteers, including African American, Caucasian, male and female participants, will be recruited from parents of patients seen in the pediatric dermatology clinic. Each participant will receive 7ml of broccoli sprout extract (BSE) in jojoba oil, containing 3500nmol of sulforaphane (Please see the preparation of broccoli sprout extract below). 500nmol of sulforaphane will be applied each night. The participants will apply the BSE-jojoba oil mixture over a circle, 3cm in diameter, on the upper arm every night for 7 consecutive nights. The control arm will have only jojoba oil applied. Both arms will be occluded with saran wrap every night. After the seventh night, the volunteers will have a 6mm biopsy taken from each arm (2 total), performed by a dermatology resident. The biopsies will be cleaned with alcohol, numbed with 0.5-1cc of 1% lidocaine with epinephrine, and closed with one 4-0 nylon nonabsorbable suture. The biopsy site will be covered with Vaseline and a bandaid. The area will be kept covered for 24 hours, after which it may be washed with soap and water and then recovered with Vaseline and a bandaid. The suture will be removed 10-14 days after the procedure. From the initial visit through the final visit for suture removal, we expect the duration of the trial to last approximately 1 month. The participants will be told to avoid applying any topical medications or over the counter lotions or creams for the duration of the study and will also be told to wash with Dove soap in the shower. They will also be advised to avoid a diet high in cruciferous plants such as broccoli, mustard, and horseradish. The biopsy results will each be divided in half. One half to be frozen for cryosectioning and immunofluorescence staining and the other half to be used for protein or RNA extraction for molecular assays (real time polymerase chain reaction and/or quantitative polymerase chain reaction for select messenger RNAs and western blotting for select protein antigens). The levels of keratin 1, keratin 5, keratin 10, keratin 14, keratin 16, keratin 17, and Nrf2 will be studied with both immunofluorescence and RNA PCR.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend 3 visits at the designated times.

Exclusion Criteria:

* Pregnant
* Known allergy to broccoli, lidocaine, or epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Immunohistochemistry | Within 1 month of skin biopsy
  Immunohistochemistry of protein levels of keratin 1, keratin 5, keratin 10, keratin 14, keratin 16, keratin 17, and Nrf2
Real time- Polymerase Chain Reaction | Within 1 month of skin biopsy
  Real time- Polymerase Chain Reaction of protein levels of keratin 1, keratin 5, keratin 10, keratin 14, keratin 16, keratin 17, and Nrf2

SECONDARY OUTCOMES:
Adverse Events | During the trial until 2 months after the trial ends
  Any adverse events associated with topical application of the drug or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cohen, MD, Principal Investigator — Professor of Dermatology
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States